CLINICAL TRIAL: NCT07054164
Title: Effects of Dual-Task Aerobic Exercise Training on Attention, Balance, and Quality of Life in Children With Specific Learning Disorder
Brief Title: Effect of Dual-Task Aerobic Exercise on Children With Specific Learning Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Mehmet Hakan Özdemir, Professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BVU-FTR-HRC-01
Record Dates: First submitted 2025-06-16; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Specific Learning Disorder
Keywords: Specific Learning Disorder; Aerobic Exercise
MeSH Terms: conditions — Specific Learning Disorder | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants were divided into three groups: a dual-task aerobic exercise group, an aerobic exercise group, and a control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment will be performed by a investigator who was blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dual-task aerobic exercise group (Other): 3 days a week, 50 minutes (10 warm-ups, 30 minutes of moderate-high intensity walking, 10 minutes of cooling down) moderate-high intensity treadmill aerobic training was provided under the supervision of a physiotherapist. In addition to aerobic training, some cognitive tasks were given to the participants during the treadmill walks.
  Interventions: Other: dual-task aerobic exercise
- aerobic exercise group (Other): 3 days a week, 50 minutes (10 warm-ups, 30 minutes of moderate-high intensity walking, 10 minutes of cooling down) moderate-high intensity treadmill aerobic training was provided under the supervision of a physiotherapist.
  Interventions: Other: aerobic exercise
- control group (No Intervention): no intervention

INTERVENTIONS:
Other: dual-task aerobic exercise — In addition to aerobic training during treadmill walks, participants were given some cognitive tasks and were asked to continue these tasks throughout the exercise.
  Arms: dual-task aerobic exercise group
Other: aerobic exercise — Aerobic training with a treadmill at medium-high intensity, 3 days a week, for 8 weeks, accompanied by a physiotherapist
  Arms: aerobic exercise group

SUMMARY:
The aim of the present study is to investigate the effects of dual-task aerobic exercise training on attention, balance, and quality of life in children with Specific Learning Disorder.

DETAILED DESCRIPTION:
Specific Learning Disorder is a neurodevelopmental condition characterized by difficulties in basic academic skills such as reading, writing, language comprehension, mathematical calculations, and information processing, despite normal or above-normal intellectual capacity.

Although the primary difficulties experienced by individuals diagnosed with Specific Learning Disorder involve impairments in acquiring academic skills such as learning and performing mathematical calculations, various deficiencies have also been observed in physical domains such as balance and motor coordination.

No previous studies have been identified in the literature examining the effects of dual-task focused aerobic exercises on individuals diagnosed with Specific Learning Disorder. The investigators hypothesize that dual-task focused aerobic exercise training administered to children with Specific Learning Disorder will have positive effects on attention, balance, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a specific learning disorder according to DSM-V criteria
* Being between the ages of 6-14
* Having reading skills
* Not having received treatment for a specific learning disorder

Exclusion Criteria:

* Having a chronic and serious systemic disease
* Having a seizure-like neurological disorder
* Having vision, speech and hearing problems
* Not attending the individual education program regularly
* Having any contraindications for physical exercise

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Stroop Test TBAG Form | 8 weeks
  The Stroop Test TBAG Form is a neuropsychological test that evaluates complex attention, focused and selective attention, resistance to disruptive stimuli, cognitive inhibition, information processing speed and executive functions.
  Unit of Measure: Points

SECONDARY OUTCOMES:
Pediatric Balance Scale (PDS) | 8 weeks
  The scale consists of 14 sections in total and each section is evaluated and scored between 0-4 points. The total score gives the PDS score. The score range of the scale is between 0-56 and higher scores indicate better balance performance.
Biodex Balance System | 8 weeks
  The Biodex Balance System is an equipment that can be used for both objective assessment of postural balance and balance training. The device consists of a screen, a circular balance platform, arm support and a printer.
Quality of Life Inventory for Children (PedsQL) | 8 weeks
  It is a scale used to evaluate the general quality of life of children aged 2-18; it consists of a total of 23 items that question children's physical, emotional, psychosocial and school-related problems, and each item is scored between 0-100.
Body composition measurement | 8 weeks
  The Omron BF511 Body Composition Monitor® non-invasive body composition measurement device, which works with the 4-pole bioelectrical impedance method (determines the ratio of fat and muscle tissue in the body with a weak electric current passing through the body), was used to calculate the participants' skeletal muscle mass ratio (%), body fat ratio (%) and basal metabolic rate.
Body Weight Measurement | 8 weeks
  Body weight will be measured using a digital scale with participants wearing light clothing and no shoes.
  Unit of Measure: Kilograms (kg)
Height Measurement | 8 weeks
  Height will be measured using a stadiometer with participants standing upright without shoes, heels together, and head in the Frankfurt plane.
  Unit of Measure: Meters (m)
Body Mass Index (BMI) | 8 weeks
  BMI will be calculated using the formula: weight in kilograms divided by the square of height in meters (kg/m²).
  Unit of Measure: Kilograms per square meter (kg/m²)

CONTACTS AND LOCATIONS:
Overall Officials: Elif DURGUT, Assistant Professor, Ph.D., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, TR, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No